CLINICAL TRIAL: NCT02949167
Title: MyHealth: Nurse-led Compared to Physician-led Breast Cancer Follow-up: A Randomized Controlled Trial
Brief Title: MyHealth: Follow-up After Breast Cancer Treatment
Acronym: MyHealth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Danish Cancer Society (Other)
Collaborators: Region Sjælland (Other)
Responsible Party: Principal Investigator, Christoffer Johansen, Professor, Danish Cancer Society
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Record.12714019
Record Dates: First submitted 2016-10-25; First posted 2016-10-31 (Estimated); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Breast Cancer
Keywords: Nurse-led follow-up after breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MyHealth intervention arm (Experimental): Nurse-led follow-up
  Interventions: Behavioral: MyHealth
- MyHealth Control condition (No Intervention): Physician-led follow-up

INTERVENTIONS:
Behavioral: MyHealth — The MyHealth intervention is a nurse-led individually tailored symptom management program, focused on patient education and regularly collection of Patient Reported Outcomes (PRO) subsequently evaluated by specialist nurses and navigation to health care service. The nurse will meet with the patient on three-five planned appointments focused on adjustment of life after breast cancer treatment including information on symptoms of relapse or late effects and how to react on these. Close relatives are invited if patients accept. Patients will report PRO´s on symptoms of recurrence and late effects every three months during the first year and thereafter every six months.The appointments with the nurse are finalized within 3-6 month and patients will be followed with PRO for three years.
  Arms: MyHealth intervention arm

SUMMARY:
Approximately 24,000 women attend a follow-up care program after end of primary treatment for breast cancer (BC) in Denmark. There is no well-conducted, larger randomized controlled trials (RCT) outlining a gold standard for follow-up programs ensuring early detection of recurrence, good management of symptoms and cost-effectiveness. The primary aim of this randomised, controlled trial is to test whether a nurse-led individually tailored symptom management program (MyHealth) will significantly reduce reported symptoms among BC patients following primary treatment compared to physician-led scheduled follow-up. Secondary, the investigators will examine patient activation (self-management), anxiety, depression, fear of recurrence, work ability, time to recurrence, overall survival, health behavior changes, health care utilization and financial costs in the two arms.

The MyHealth program provides patients with a nurse-led education focusing on management of symptoms, an electronic platform to report symptoms to the nurses and support in symptom management and navigation of patients to appropriate health care services.

DETAILED DESCRIPTION:
During an 18-month period, 494 primary BC patients will be recruited from the Departments of Oncology at Naestved and Roskilde Hospital. The women will be enrolled in the study following completion of primary treatment. Participants are randomized 1:1 to the intervention (Nurse-led follow up) or control group (physician-led follow-up) and followed for 5 years. No matter group assignment, all women will follow the national mammography screening programs.

Patients who accept to participate are asked to invite a close relative, preferably partners, to participate in the study. Patients, who do not want to participate in the randomization will be asked if they are willing to participate in the study by filling out two questionnaires. Patients who decline to participate in the MyHealth study will be enrolled in the standard follow-up.

The investigators will collect data using questionnaires, clinical databases, and national registers before intervention and for 5 years after inclusion both in the control and intervention arm. Questionnaires from validated scales are used to measure primary and secondary outcomes in both groups whereas Patient Reported Outcomes (PRO) are only collected in the intervention group. Patients who experiences relapse during the MyHealth intervention will not be asked to fill in the remaining outcome questionnaires or PROs since they quit the follow-up program in favor of treatment for recurrent disease.

During follow-up, the patient will consult the nurse or the project physician if PROs reveal a need, or if the patient require a consultation. In order to ensure that treatment of symptoms and referral to other health professionals will meet clinical guidelines the nurses are instructed to follow a detailed response algorithm, which is developed by the project physician in collaboration with experienced oncologists.

ELIGIBILITY:
Inclusion Criteria:

* Complete remission following primary treatment for loco-regional BC (stage I-II) - No confirmed genetic predisposition to BC
* Female gender
* Performance status ≤3
* Read, understand and speak Danish
* No severe cognitive problems
* No severe psychiatric disease requiring treatment or any substance abuse.

Exclusion Criteria:

* Genetic predisposition for BC
* Patient younger than 40 years of age at diagnosis
* Control after recurrent breast cancer
* Other active cancer except non-melanoma skin cancer
* Severe cognitive problems or dementia
* Severe psychiatric disease requiring treatment, e.g. schizophrenia, alcohol or narcotic dependence

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 503 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Changes in breast cancer specific symptom burden (TOI-PFB) | at inclusion, 6 months,12 months, 24 months, 36 months and 60 months
  Trial Outcome Index-Physical/Functional/Breast (TOI-PFB) score of the Functional Assessment of Cancer Therapy -Breast (FACT-B) Domains: Physical well-being, Functional wellbeing,BC symptoms

SECONDARY OUTCOMES:
Changes in breast cancer specific symptom burden | at inclusion, 6 months,12 months, 24 months, 36 months and 60 months
  Functional Assessment of Cancer Therapy -Breast (FACT-B) Domains: Physical well-being, social/family well-being, Emotional well-being,Functional wellbeing, BC symptoms
Changes in knowledge, skill, and confidence for self-management | at inclusion, 6 months,12 months, 24 months, 36 months and 60 months
  Patient Activation Measure (PAM)
Changes in anxiety | at inclusion, 6 months,12 months, 24 months, 36 months and 60 months
  Generalized Anxiety Disorder (GAD-7)
Changes in self-management | at inclusion, 6 months,12 months, 24 months, 36 months and 60 months
  The Health Education Impact Questionnaire (heiQ)
Changes in fear of recurrence | at inclusion, 6 months,12 months, 24 months, 36 months and 60 months
  Concerns About Recurrence Questionnaire (CARQ-4)
Changes in Depression | at inclusion, 6 months,12 months, 24 months, 36 months and 60 months
  The Patient Health Questionnaire (PHQ-9)
Changes in work ability | at inclusion, 6 months,12 months, 24 months, 36 months and 60 months
  Work Ability Index (WAI)
Changes in quality-adjusted life year (QALY) | at inclusion, 6 months,12 months, 24 months, 36 months and 60 months
  EuroQol 5 domains (5D), 5 levels (5L)

OTHER OUTCOMES:
Health Care Use | at 60 months
  Study specific items on health care use single items

CONTACTS AND LOCATIONS:
Overall Officials: Christoffer Johansen, Professor, Principal Investigator — The Cancer Society Research Center, Survivorship; Mads N Svendsen, MD, PHD, Principal Investigator — The Department for Oncology Naestved and Roskilde Hospital
Locations (1):
- Department of Oncology and Palliative Care, Naestved Hospital, Næstved, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Saltbaek L, Bidstrup PE, Karlsen RV, Hoeg BL, Horsboel TA, Belmonte F, Andersen EAW, Zoffmann V, Friberg AS, Svendsen MN, Christensen HG, Glavicic V, Nielsen DL, Dalton SO, Johansen C. Nurse-Led Individualized Follow-Up Versus Regular Physician-Led Visits After Early Breast Cancer (MyHealth): A Phase III Randomized, Controlled Trial. J Clin Oncol. 2024 Jun 10;42(17):2038-2049. doi: 10.1200/JCO.23.01447. Epub 2024 Mar 18. PMID 38498781